CLINICAL TRIAL: NCT06453460
Title: Prospective Evaluation of Efficacy of CMV-specific T Cell Immunity (CMV-TCIP) Directed Letermovir Prophylaxis After Allogeneic Hematopoietic Cell Transplantation
Brief Title: CMV-TCIP Directed Letermovir Prophylaxis After Allo-SCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eurofins Viracor (Unknown)
Responsible Party: Principal Investigator, Piyanuch Kongtim, Associate Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4005; UCI 22-188 (Other: UCI)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: CMV; Allogeneic Stem Cell Transplantation
Keywords: CMV T Cell Immunity Panel; CMV reactivation; Allogeneic stem cell transplantation; Letermovir
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AHCT recipients (Experimental)
  Interventions: Drug: Letermovir; Device: CMV T Cell Immunity Panel (CMV-TCIP); Diagnostic Test: CMV DNA PCR

INTERVENTIONS:
Drug: Letermovir — Subjects will receive 14 weeks of letermovir prophylaxis at standard recommended dose follow by CMV-TCIP-directed extended prophylaxis.
Device: CMV T Cell Immunity Panel (CMV-TCIP) — Viracor CMV-TCIP assay to measure how a person's immune system responds to CMV. Viracor CMV-TCIP will be measured monthly, starting at week 14, until positive, then at week 30 and 52.
Diagnostic Test: CMV DNA PCR — Plasma level of CMV DNA PCR will be measured at enrollment and at least weekly through week 30, then at least every 2 weeks through week 52 of transplant if no GVHD or CMV reactivation.

SUMMARY:
This is a phase 2, prospective cohort clinical trial evaluating the utilization of CMV T Cell Immunity Panel (CMV-TCIP) assay to guide the duration of primary CMV prophylaxis in CMV-seropositive recipients of allogeneic stem cell transplant or recipients receiving a stem cell graft from a CMV serology positive donor.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age on the day of signing informed consent.
* Karnofsky performance >70%
* Have documented seropositivity for CMV (either donor or recipient CMV IgG seropositivity) before AHCT.
* Eligible for AHCT from an HLA-matched related, matched unrelated, mismatched unrelated or haploidentical donor using either bone marrow or peripheral blood stem cells.
* Have undetectable CMV DNA from a plasma sample collected within 5 days prior to enrollment.
* Must be within Day-10 thru Day+28 days of planned HSCT at the time of enrollment.
* Be able to comply with medical recommendations or follow-up.
* Has adequate organ functions determined by

  1. Serum creatinine clearance ≥50 ml/min (calculated with Cockroft-Gault formula).
  2. Bilirubin ≤1.5 mg/dl except for Gilbert's disease.
  3. ALT or AST ≤200 IU/ml for adults.
  4. Conjugated (direct) bilirubin < 2x upper limit of normal.
  5. Left ventricular ejection fraction ≥40%.
  6. Diffusing capacity for carbon monoxide (DLCO) ≥ 50% predicted corrected for hemoglobin.

Exclusion Criteria:

* Has a history of CMV end-organ disease or CS-CMVi within 6 months prior to enrollment.
* Received within 7 days prior to screening or plans to receive during the study any of the following:

  1. Ganciclovir
  2. Valganciclovir
  3. Foscarnet
  4. Acyclovir (> 3200 mg PO per day or > 25 mg/kg IV per day)
  5. Valacyclovir (> 3000 mg/day)
  6. Famciclovir (> 1500 mg/day)
* Received within 30 days prior to screening or plans to receive during the study any of the following drugs: cidofovir, CMV hyper-immune globulin, any investigational CMV antiviral agent/biologic therapy.
* Has suspected or known hypersensitivity to active or inactive ingredients of letermovir formulations.
* Has an uncontrolled infection
* Requires mechanical ventilation or is hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinically significant cytomegalovirus infection (CS-CMVi) at 52 weeks after transplant | 1 year after transplant
  Number of patients who develop CS-CMVi within 52 weeks after receiving a transplant

SECONDARY OUTCOMES:
Cumulative incidence of CMV disease at 52 weeks after transplant | 1 year after transplant
  Number of patients who develop CMV disease within 52 weeks after receiving a transplant
Cumulative incidence of CMV related death at 52 weeks | 1 year after transplant
  Number of patients who die from complications directly attributable to CMV infection within 52 weeks
Overall Survival at 1 year after transplant | 1 year after transplant
  Number of patients who survive beyond 1 year after transplant
Positive predictive value of CMV-TCIP assay after transplant in predicting CS-CMVi protection | 1 year after transplant
  Positive predictive value of CMV-TCIP assay at 14 weeks after transplant in predicting CS-CMVi protection through 1 year after transplant in patients who had letermovir discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Piyanuch Kongtim, MD,PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No